CLINICAL TRIAL: NCT02213588
Title: Effects of Plant Concentrate Blend on Oxidative Stress in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABG AOX-2 Efficacy
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Antioxidant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AOX blend (Active Comparator): Rosemary:Quercetin:Turmeric (300 mg total)
  Interventions: Dietary Supplement: AOX blend
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AOX blend — Antioxidant supplement
  Other Names: Antioxidant blend
  Arms: AOX blend
Dietary Supplement: Placebo
  Other Names: Placebo sugar pill
  Arms: Placebo

SUMMARY:
This study evaluates the response to oxidative stress in healthy men and women after taking a blend of plant concentrate.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how blends of plant concentrates impacts oxidative stress in humans. Biomarkers of oxidative stress will be measured at three time points in 3 month intervention. Based on our proof of concept dose response study, it was shown that the plant concentrate at the proposed dose can lower markers of oxidative damage and induce the production of antioxidant enzymes. We would like to confirm these findings and further evaluate the implication of increased antioxidative enzymes as seeing in our proof of concept study. An acute oxidative stress will be induced by a high glycemic drink and short aerobic exercise and the response during the induction of an acute oxidative stress as well as the recovery from an acute oxidative stress. Since the induction of antioxidative enzymes not only is linked to the protection of proteins and lipids from oxidative damage, it is also linked to the protection of DNA damage. Therefore, in this study, comet assay will be performed to evaluate the integrity of DNA.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women between 18 - 65 yr with low fruit and vegetable intake.
2. Individual with low fruit and vegetable intake and consuming fewer than 12 items found on the Recommended Foods Checklist (RFC) (APPENDIX I) per week. (score < 12 points
3. Safety data: Blood chemistry results specifically Blood Urea Nitrogen (BUN), Serum Creatinine, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-glutamyl transpeptidase (GGTP), Total Bilirubin and alkaline phosphatase and urinalysis results, specifically urine pH, protein, glucose, ketone and bilirubin levels within +/- 20% of normal value indicated in the lab report.
4. Subjects with laboratory test results exceeding by >20% of the upper limit of the reference range in Creatine Phosphokinase, uric acid or blood glucose may be included in the study if the Principal Investigator decides those subjects are sufficiently healthy to participate safely in the study.
5. Individual should be judged to be in good general health on the basis of an interview and a physician will perform an abbreviated physical exam.
6. Individual understands the procedures and agrees to participate in the study.
7. Individual is willing to maintain their exercise habits and dietary pattern throughout the duration of the trial except as instructed to avoid high content of quercetin (for example, quercetin can be found in apple and onion), rosemary, turmeric throughout the duration of the trial.
8. Individual is willing to consume a diet or drinks devoid with high content of quercetin (for example, quercetin can be found in apple and onion), rosemary, turmeric throughout the duration of the trial.
9. Individual is able and willing to provide written informed consent and confidentiality agreement.

Exclusion Criteria:

* Persons will be excused from participating in the study if any of the following conditions exist:

  1. Use of dietary supplements within one week of Day 1. Supplements include any vitamins, minerals, and herbal products, including herbal drinks.
  2. Presence of, or clinical significant history of, cancer, cardiovascular, endocrine, kidney, liver, lung, gastrointestinal, metabolic disorder, absorption disorder such as Celiac or Crohn's disease and/or any other chronic health condition such as diabetes identified from the findings of the interview.
  3. Presence of gallstones or history of gallbladder disease.
  4. Presence or history of diabetes.
  5. Presence of cardiovascular disease and hypertension with inconsistent medication regimen, unstable conditions, and without proper physician's supervision identified from the findings of the interview.
  6. Ten hours prior to the blood and urine sample collection, subjects should refrain from using medications such as statins (e.g., simvastatin, fluvastatin), NSAIDS including aspirin, nitric oxide (eNOS) activators or inhibitors (e.g., selegiline, Viagra), and angiotensin II receptor blocker (e.g., Telmisartan (blood pressure)), take any of these medications Participant who eats spicy food (e.g., capsaicin from chili pepper) and/or drinks coffee and teas including herbal teas within 10 hours prior to the blood and urine sample collection.
  7. Participation in another clinical trial within 30 days of enrollment into the study.
  8. History or current abuse of nicotine, drugs or alcohol, or intake > 3 alcoholic beverages per day
  9. Have known allergy to the ingredients in the tested samples such as quercetin, rosemary, turmeric, Holy basil, wasabi, broccoli seed, and licorice.
  10. Any condition that the Principal Investigator believes may put the subject at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in urine isoprostane | Baseline, 3 mo
  Change from baseline in urinary antioxidant biomarker in 3 months.

SECONDARY OUTCOMES:
Change in plasma isoprostane | baseline, 3 mo
  Change in baseline blood antioxidant marker from baseline to 3 month
Change in erythrocyte lysate superoxide dismutase | baseline, 3.0 mo
  Change in antioxidant biomarker from baseline to 3 months
Change in plasma superoxide dismutase | baseline, 3.0 mo
  Change in antioxidant biomarker from baseline to 3 months
Change in plasma catalase | baseline, 3.0 mo
  Change in antioxidant biomarker from baseline to 3 months
Change in plasma 3-nitrotyrosine | baseline, 3.0 mo
  Change in antioxidant biomarker from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Keech, M.D., Principal Investigator — Southbay Pharma Research
Locations (1):
- Southbay Pharma Research, Buena Park, California, United States